CLINICAL TRIAL: NCT02455518
Title: Comparative Efficacy of 4 Oral Analgesics for the Initial Management of Acute Musculoskeletal Extremity Pain
Brief Title: Comparative Efficacy of 4 Oral Analgesics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Andrew Chang, MD, PI, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-4156
Record Dates: First submitted 2015-05-22; First posted 2015-05-28 (Estimated); Results first posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain | interventions — oxycodone-acetaminophen; acetaminophen, codeine drug combination; Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Oxycodone/acetaminophen (Active Comparator): Oxycodone/acetaminophen (5 mg/325 mg)
  Interventions: Drug: Oxycodone/acetaminophen
- Hydrocodone/acetaminophen (Active Comparator): Hydrocodone/acetaminophen (5 mg/300 mg)
  Interventions: Drug: Hydrocodone/acetaminophen
- Codeine/acetaminophen (Active Comparator): Codeine/acetaminophen (30 mg/300 mg)
  Interventions: Drug: Codeine/acetaminophen
- Ibuprofen/acetaminophen (Active Comparator): Ibuprofen/acetaminophen (400 mg/1000 mg)
  Interventions: Drug: Ibuprofen/acetaminophen

INTERVENTIONS:
Drug: Oxycodone/acetaminophen
  Other Names: Percocet
  Arms: Oxycodone/acetaminophen
Drug: Hydrocodone/acetaminophen
  Other Names: Norco
  Arms: Hydrocodone/acetaminophen
Drug: Codeine/acetaminophen
  Other Names: Tylenol with codeine
  Arms: Codeine/acetaminophen
Drug: Ibuprofen/acetaminophen
  Arms: Ibuprofen/acetaminophen

SUMMARY:
The purpose of this study is to perform a randomized, double blind 4-arm clinical trial of the comparative efficacy of 4 oral analgesics in the initial management of acute musculoskeletal extremity pain presenting to the ED.

DETAILED DESCRIPTION:
To perform a randomized, double blind 4-arm clinical trial of the comparative efficacy of 4 oral analgesics in the initial management of acute musculoskeletal extremity pain presenting to the ED. The 4 groups are as follows:

1. Oxycodone/acetaminophen (5/325)
2. Hydrocodone/acetaminophen (5/325)
3. Codeine/acetaminophen (30/300)
4. Ibuprofen/acetaminophen (400/1000)

ELIGIBILITY:
Inclusion Criteria:

* Complaint of acute pain of < 7 days duration
* Location of pain in one or more extremities defined as distal to and including the shoulder joint in the upper extremities and distal to and including the hip joint in the lower extremities;
* Radiologic evaluation is planned

Exclusion Criteria:

* Inability to confirm reliable means of phone followup.
* Past use of methadone
* Chronic condition requiring frequent pain management such as sickle cell disease, fibromyalgia, or any neuropathy
* History of an adverse reaction to any of the study medications
* Opioids taken in the past 24 hours
* Ibuprofen or acetaminophen taken in past 8 hours
* Pregnancy by either urine or serum HCG testing
* Breastfeeding per patient report
* History of peptic ulcer disease
* Report of any prior use of recreational narcotics
* Medical condition that might affect metabolism of opioid analgesics, acetaminophen, or ibuprofen such as hepatitis, renal insufficiency, hypo- or hyperthyroidism, Addison's or Cushing's disease
* Taking any medicine that might interact with one of the study medications, such as antidepressant SSRI's or Tricyclics, antipsychotics, anti-malaria medications quinidine or halofantrine, Amiodarone or Dronedarone, diphenhydramine, celecoxib, ranitidine, cimetidine, ritanovir, terbinafine, or St John's Wort.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2017-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Chang AK, Bijur PE, Esses D, Barnaby DP, Baer J. Effect of a Single Dose of Oral Opioid and Nonopioid Analgesics on Acute Extremity Pain in the Emergency Department: A Randomized Clinical Trial. JAMA. 2017 Nov 7;318(17):1661-1667. doi: 10.1001/jama.2017.16190. PMID 29114833

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxycodone/Acetaminophen: Oxycodone/acetaminophen (5 mg/325 mg)
  Oxycodone/acetaminophen
- Hydrocodone/Acetaminophen: Hydrocodone/acetaminophen (5 mg/300 mg)
  Hydrocodone/acetaminophen
- Codeine/Acetaminophen: Codeine/acetaminophen (30 mg/300 mg)
  Codeine/acetaminophen
- Ibuprofen/Acetaminophen: Ibuprofen/acetaminophen (400 mg/1000 mg)
  Ibuprofen/acetaminophen
Period: Overall Study
Arm/Group | Oxycodone/Acetaminophen | Hydrocodone/Acetaminophen | Codeine/Acetaminophen | Ibuprofen/Acetaminophen
Started | 104 | 104 | 104 | 104
Completed | 104 | 103 | 103 | 101
Not Completed | 0 | 1 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone/Acetaminophen | Hydrocodone/Acetaminophen | Codeine/Acetaminophen | Ibuprofen/Acetaminophen | Total
Number analyzed (Participants) | 104 | 103 | 103 | 101 | 411
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (12) | 37 (13) | 37 (12) | 37 (11) | 37 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 44 | 54 | 199
  Male | 54 | 52 | 59 | 47 | 212
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latino | 62 | 65 | 58 | 62 | 247
  African-American | 29 | 26 | 33 | 34 | 122
  Caucasian | 7 | 8 | 6 | 2 | 23
  East Asian/Asian | 2 | 3 | 3 | 3 | 11
  Other | 4 | 1 | 3 | 0 | 8
Region of Enrollment [Number; unit: participants]
  United States | 104 | 103 | 103 | 101 | 411

OUTCOME MEASURES:

1. Primary Outcome: Between Group Difference in Change in Numerical Rating Scale (NRS) Pain Scores
Description: Change in numerical rating scale (NRS) pre and 2 hours post receiving study medication while in the ED. The NRS is a validated 11-point numerical scale that ranges from 0 (no pain) to 10 (worst pain possible)
Time Frame: 2 hours
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Oxycodone/Acetaminophen | Hydrocodone/Acetaminophen | Codeine/Acetaminophen | Ibuprofen/Acetaminophen
Number analyzed (Participants) | 104 | 103 | 103 | 101
units on a scale | 4.4 [3.7 to 5.0] | 3.5 [2.9 to 4.2] | 3.9 [3.2 to 4.5] | 4.3 [3.6 to 4.9]

2. Secondary Outcome: Between Group Difference in Change in Numerical Rating Scale (NRS) Pain Scores
Description: Change in numerical rating scale (NRS) pre and 1-hour post receiving study medication while in the ED. The NRS is a validated 11-point numerical scale that ranges from 0 (no pain) to 10 (worst pain possible)
Time Frame: 1 hour
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Oxycodone/Acetaminophen | Hydrocodone/Acetaminophen | Codeine/Acetaminophen | Ibuprofen/Acetaminophen
Number analyzed (Participants) | 104 | 103 | 103 | 101
units on a scale | 3.1 [2.6 to 3.7] | 2.4 [1.8 to 3.0] | 2.7 [2.1 to 3.3] | 2.9 [2.4 to 3.5]

ADVERSE EVENTS:
Time Frame: Adverse events were not collected
Arm/Group | Oxycodone/Acetaminophen | Hydrocodone/Acetaminophen | Codeine/Acetaminophen | Ibuprofen/Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT02455518/Prot_SAP_000.pdf
  • Informed Consent Form (2015-05-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT02455518/ICF_001.pdf